CLINICAL TRIAL: NCT00607074
Title: Effects of Anti-Giardia and Antihelmintic Treatment on Infant Nutritional and Biochemical Status and Intestinal Permeability in Rural Bangladesh
Brief Title: Impact of Anti-Giardia and Antihelmintic Treatment on Infant Growth in Bangladesh
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Cambridge (Other)
Responsible Party: Dr Rie Goto, Department of Biological Anthropology, University of Cambridge
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BMRC/ERC/2001-2004/2281; BMRC/ERC/2001-2004/2281
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2008-02-05 (Estimated); Status verified 2008-01

CONDITIONS: Giardiasis
MeSH Terms: conditions — Giardiasis | interventions — secnidazole; Albendazole; Control Groups

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: Anti-Giardia and antihelmintic treatment (secnidazole or albendazole); Drug: Anti-Giardia treatment only (secnidazole or albendazole); Drug: Control group (placebo)

INTERVENTIONS:
Drug: Anti-Giardia and antihelmintic treatment (secnidazole or albendazole) — Every 4 weeks: Secnidazole (70mg/ml suspension, 0.5ml per kg of body weight) or a placebo was administered Every 12 weeks: Albendazole (syrup, 200mg)
Drug: Anti-Giardia treatment only (secnidazole or albendazole) — Every 4 weeks: Secnidazole (70mg/ml suspension, 0.5ml per kg of body weight) Every 12 weeks: placebo of Albendazole
Drug: Control group (placebo) — Every 4 weeks: Secnidazole placebo Every 12 weeks: Albendazole placebo

SUMMARY:
This longitudinal study aimed to assess whether regular anti-Giardia and antihelmintic treatment improved growth and small intestinal mucosal function of rural Bangladeshi infants.

DETAILED DESCRIPTION:
A randomised double-blind controlled intervention of 36 weeks duration was conducted in a rural community located 40kms north-west of Dhaka, the capital of Bangladesh. Infants aged between 3 and 11 months were randomly assigned to either receiving anti-Giardia and antihelmintic treatment, or anti-Giardia treatment only, or a control group receiving placebos. Weight and supine length were recorded every 4 weeks. Every 12 weeks intestinal permeability (L/M ratio), haemoglobin, plasma albumin, alpha-1-acid glycoprotein, immunoglobulin G and Giardia intestinalis specific IgM titre (GSIgM) and eggs of the three common geohelminths and Giardia intestinalis cysts were determined.

ELIGIBILITY:
Inclusion Criteria:

* infants living in the study area

Ages: 3 Months to 15 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 410 (Actual)
Dates: Start 2003-06; Primary Completion 2004-04 (Actual); Study Completion 2006-12 (Actual)

PRIMARY OUTCOMES:
nutritional status | 9 months

SECONDARY OUTCOMES:
intestinal permeability | 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas C Mascie-Taylor, ScD, Study Chair — Department of Biological Anthropology, University of Cambridge
Locations (1):
- National Institute of Preventive and Social Medicine, Mohakhali, Dhaka Division, Bangladesh

REFERENCES:
- [Derived] Goto R, Mascie-Taylor CG, Lunn PG. Impact of anti-Giardia and anthelminthic treatment on infant growth and intestinal permeability in rural Bangladesh: a randomised double-blind controlled study. Trans R Soc Trop Med Hyg. 2009 May;103(5):520-9. doi: 10.1016/j.trstmh.2008.07.020. Epub 2008 Sep 11. PMID 18789466